CLINICAL TRIAL: NCT01164488
Title: A Two-Way Interaction Study Between RO5190591/RTV and Ketoconazole in Healthy Subjects
Brief Title: A Study of RO5190591 (Danoprevir) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP25293
Record Dates: First submitted 2010-07-15; First posted 2010-07-16 (Estimated); Last update posted 2016-08-29 (Estimated); Status verified 2016-08

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — danoprevir; Ketoconazole; Ritonavir

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: danoprevir; Drug: ketoconazole; Drug: ritonavir

INTERVENTIONS:
Drug: danoprevir — Repeated daily doses
Drug: ketoconazole — Repeated daily doses
Drug: ritonavir — Repeated daily doses

SUMMARY:
This non-randomized, open-label study will evaluate the interaction of RO5190591(danoprevir)/ritonavir with and without ketoconazole and the safety and tolerability in healthy volunteers. Participants will be administered repeated daily doses of ketoconazole alone, RO5190591/ritonavir, and RO5190591/ritonavir plus ketoconazole. The anticipated time on study treatment is 25 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy volunteers, aged 18-64 years, inclusively
* Weight >/=50.0 kg
* Body Mass Index (BMI) 18.0-32.0 kg/m2
* Ability and willingness to abstain from alcohol, xanthine-containing beverages or food (coffee, tea, cola, chocolate, "energy drinks") from 48 hours prior to entry in the clinical study center until discharge
* Ability and willingness to abstain from grapefruit or grapefruit juice, star fruit, and Seville oranges from 7 days prior to entry in the clinical study center until discharge
* Medical history without major recent or ongoing pathology

Exclusion Criteria:

* Pregnant or lactating women and male partners of women who are pregnant or lactating
* Sustained supine systolic blood pressure >140 or <90 mmHG and supine diastolic blood pressure >90 or <50 mmHG at Screening or Day -1
* Resting heart rate >100 or <45 beats per minute at Screening or Day -1
* Any history of clinically significant cardiovascular or cerebrovascular disease
* Positive drug test result at screening or each admission
* Donation or loss of blood over 450 ml (1 pint) within 60 days prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To investigate the interaction between RO5190591/ritonavir and ketoconazole | Day 40

SECONDARY OUTCOMES:
To assess the safety and tolerability of multiple doses of RO5190591/ritonavir without and with ketoconazole | Day 40

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States